CLINICAL TRIAL: NCT05215990
Title: Efficacy of Metformin for Sputum Conversion in Patients With Active Pulmonary Tuberculosis: A Randomized Controlled Trial
Brief Title: Efficacy of Metformin for Sputum Conversion in Patients With Active Pulmonary Tuberculosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Principal Investigator, Angsana Phuphuakrat, Principal investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MURA2021/816
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Tuberculosis, Pulmonary
Keywords: Tuberculosis; Metformin
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — Metformin; Tablets

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient receive metformin with pulmonary tuberculosis standard treatment. (Active Comparator): Patient receive pulmonary tuberculosis standard treatment: isoniazid, rifampicin, pyrazinamide, and ethambutol in first and second month(weight adjusted dose), then in third to sixth month switch tuberculosis standard treatment to isoniazid and rifampicin(weight adjusted dose). In all 6 months, patient receive metformin (500 mg) 1 tablet simultaneously.
  Interventions: Drug: MetFORMIN 500 Mg Oral Tablet
- Patient receive placebo drug with pulmonary tuberculosis standard treatment. (Placebo Comparator): Patient receive pulmonary tuberculosis standard treatment: isoniazid, rifampicin, pyrazinamide, and ethambutol in first and second month(weight adjusted dose), then in third to sixth month switch tuberculosis standard treatment to isoniazid and rifampicin(weight adjusted dose). In all 6 months, patient receive placebo drug 1 tablet simultaneously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MetFORMIN 500 Mg Oral Tablet — studying about acid-fast bacillus sputum conversion ratio from positive to negative of pulmonary tuberculosis patients receive metformin with pulmonary tuberculosis standard treatment group in second week, second, fifth, and sixth month.
  Arms: Patient receive metformin with pulmonary tuberculosis standard treatment.
Drug: Placebo — studying about acid-fast bacillus sputum conversion ratio from positive to negative of pulmonary tuberculosis patients receive placebo drug with pulmonary tuberculosis standard treatment group in second week, second, fifth, and sixth month.
  Arms: Patient receive placebo drug with pulmonary tuberculosis standard treatment.

SUMMARY:
This study was a randomized controlled trial studying about acid-fast bacillus sputum conversion ratio from positive to negative of pulmonary tuberculosis patients between metformin with pulmonary tuberculosis standard treatment group and placebo drug with pulmonary tuberculosis standard treatment.

DETAILED DESCRIPTION:
1. Pulmonary tuberculosis Patients with presence of at least one acid-fast bacillus in the sputum will be examined by an internist.
2. Collect the necessary basic information of patients who agree to participate in the treatment such as complete blood count, blood urea nitrogen, creatinine, liver function test, fasting plasma glucose, hemoglobinA1C, lactate, and gene expression signature for tuberculosis.
3. Patients will be randomized into 2 groups: those who will receive metformin with pulmonary tuberculosis standard treatment and those who will receive placebo drug with pulmonary tuberculosis standard treatment.
4. Patients will get a chest x-ray and collect sputum acid fast bacillus, sputum culture for tuberculosis and collect blood sample laboratory such as complete blood count, liver function test, creatinine, fasting plasma glucose, lactate, and gene expression signature for tuberculosis at second week.
5. Patients will get a chest x-ray and collect sputum acid fast bacillus, and sputum culture for tuberculosis at second month.
6. Patients will get a chest x-ray and collect sputum acid fast bacillus, and sputum culture for tuberculosis at fifth month.
7. Patients will get a chest x-ray and collect sputum acid fast bacillus, and sputum culture for tuberculosis at sixth month.
8. After collecting all information of patients, Investigators will analyze in clinical and statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old
* Be diagnosed pulmonary tuberculosis compatible with clinical and chest x ray by an internist
* Presence of at least one acid -fast bacillus in the sputum
* Recieve pulmonary tuberculosis standard treatment compose of isoniazid, rifampicin, pyrazinamide and ethambutol
* BMI more than 18.5 kg/m2
* Reserach participants were diagnosed diabetes or non diabetes.
* Research participants or representatives are welcome to join the project by signing.

Exclusion Criteria:

* Pregnancy
* Organ transplants
* eGFR less than 45 ml/min/1.73 m2
* AST, ALT or total bilirubin more than three times
* Researh participants have received metformin at least 2 weeks before joining the project.
* Immunocompromised host such as patient receive systemic immunosuppressive drugs or systemic chemotherapy.
* Research participant or his representative refuses or requests to withdraw,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
To study about acid-fast bacillus sputum conversion ratio from positive to negative of pulmonary tuberculosis patients between metformin and placebo drug with pulmonary tuberculosis standard treatment. | 6 months
  patient will be collected sputum acid fast bacillus and sputum culture for tuberculosis in second week, second, fifth, sixth month.

SECONDARY OUTCOMES:
To study about side effect such as nausea, vomit, hepatitis between patients use metformin with pulmonary tuberculosis standard treatment and patients use placebo drug with pulmonary tuberculosis standard treatment. | 6 months
  To compare incidence rate of side effect between patients use metformin with pulmonary tuberculosis standard treatment and patients use placebo drug with pulmonary tuberculosis standard treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Angsana Phuphuakrat, Ratchathewi, ฺBangkok, Thailand

REFERENCES:
- [Background] Singhal A, Jie L, Kumar P, Hong GS, Leow MK, Paleja B, Tsenova L, Kurepina N, Chen J, Zolezzi F, Kreiswirth B, Poidinger M, Chee C, Kaplan G, Wang YT, De Libero G. Metformin as adjunct antituberculosis therapy. Sci Transl Med. 2014 Nov 19;6(263):263ra159. doi: 10.1126/scitranslmed.3009885. PMID 25411472
- [Background] Lee YJ, Han SK, Park JH, Lee JK, Kim DK, Chung HS, Heo EY. The effect of metformin on culture conversion in tuberculosis patients with diabetes mellitus. Korean J Intern Med. 2018 Sep;33(5):933-940. doi: 10.3904/kjim.2017.249. Epub 2018 Mar 16. PMID 29540054
- [Background] Degner NR, Wang JY, Golub JE, Karakousis PC. Metformin Use Reverses the Increased Mortality Associated With Diabetes Mellitus During Tuberculosis Treatment. Clin Infect Dis. 2018 Jan 6;66(2):198-205. doi: 10.1093/cid/cix819. PMID 29325084
- [Background] Yu X, Li L, Xia L, Feng X, Chen F, Cao S, Wei X. Impact of metformin on the risk and treatment outcomes of tuberculosis in diabetics: a systematic review. BMC Infect Dis. 2019 Oct 17;19(1):859. doi: 10.1186/s12879-019-4548-4. PMID 31623569
- [Background] Lashen H. Role of metformin in the management of polycystic ovary syndrome. Ther Adv Endocrinol Metab. 2010 Jun;1(3):117-28. doi: 10.1177/2042018810380215. PMID 23148156
- [Background] Ning HH, Le J, Wang Q, Young CA, Deng B, Gao PX, Zhang HQ, Qin SL. The effects of metformin on simple obesity: a meta-analysis. Endocrine. 2018 Dec;62(3):528-534. doi: 10.1007/s12020-018-1717-y. Epub 2018 Aug 27. PMID 30151735
- [Background] Novita BD, Ali M, Pranoto A, Soediono EI, Mertaniasih NM. Metformin induced autophagy in diabetes mellitus - Tuberculosis co-infection patients: A case study. Indian J Tuberc. 2019 Jan;66(1):64-69. doi: 10.1016/j.ijtb.2018.04.003. Epub 2018 Apr 17. PMID 30797286
- [Result] Vashisht R, Brahmachari SK. Metformin as a potential combination therapy with existing front-line antibiotics for Tuberculosis. J Transl Med. 2015 Mar 7;13:83. doi: 10.1186/s12967-015-0443-y. PMID 25880846
- See also: Clinical Evaluation of Efficacy and Safety of Metformin add-on Therapy to Standard ATT in Newly Diagnosed Pulmonary Tuberculosis Patients — https://biomedpharmajournal.org/vol13no1/clinical-evaluation-of-efficacy-and-safety-of-metformin-add-on-therapy-to-standard-att-in-newly-diagnosed-pulmonary-tuberculosis-patients/